CLINICAL TRIAL: NCT06725628
Title: Multiomics Study of Biological Behavior of Lymph Node Metastasis in Papillary Thyroid Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Tianhan Zhou (Other Government)
Responsible Party: Sponsor-Investigator, Tianhan Zhou, Clinical Professor, Zhejiang Chinese Medical University
Organization: Zhejiang Chinese Medical University (Other Government)
Other Study IDs: 2022KY153-CX1; 2022ZA119 (Other Grant/Funding Number: Huang Hai)
Record Dates: First submitted 2024-11-22; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Papillary Thyroid Carcinoma; Lymph Node Cancer Metastatic
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LNM group and NLNM group: The primary objective of this study is to evaluate the accuracy of the ThyMPR-CLNM model in predicting central lymph node metastasis (CLNM) in patients with stage T1 papillary thyroid carcinoma (PTC).
  Interventions: Diagnostic Test: Thy_CLNM_multi_omics

INTERVENTIONS:
Diagnostic Test: Thy_CLNM_multi_omics — Surgery

SUMMARY:
Establish a predictive model for assessing neck lymph node metastasis of papillary thyroid carcinoma based on metabolomics, proteomics, and imaging omics data, exploring an ideal protocal for the precise diagnosis and treatment of papillary thyroid carcinoma."

DETAILED DESCRIPTION:
This study is a multicenter, observational cohort study aimed at assessing the accuracy and effectiveness of the ThyMPR-CLNM multi-omics model in predicting CLNM in patients diagnosed with stage T1 PTC. The design incorporates the following critical components:

The study enrolled 2000 patients diagnosed with stage T1 PTC from Hangzhou Traditional Chinese Medical Hospital, affiliated with Zhejiang Chinese Medical University, between Dec.2024 and Dec.2026. Fresh frozen tumor tissue, serum samples, and preoperative ultrasound images were collected from participants. These samples were utilized for comprehensive multi-omics analyses, including metabolomic and proteomic profiling, as well as ultrasound radiomic feature extraction. To minimize selection bias and balance covariates, propensity score matching was performed in two rounds, establishing a discovery set and a validation set with matched groups based on the propensity scores calculated through logistic regression. This ensured comparable groups for subsequent analyses. The study involved analyzing the collected samples through advanced techniques such as liquid chromatography-mass spectrometry (LC-MS) for metabolomic and proteomic analyses, and Pyradiomics for extracting radiomics features from ultrasound images. Differentially expressed metabolites, proteins, and radiomic features were identified and integrated for the development of the ThyMPR-CLNM prediction model. The Least Absolute Shrinkage and Selection Operator (LASSO) regression technique was utilized to construct the ThyMPR-CLNM model based on identified features from the multi-omics analyses. The model's performance was subsequently validated using an independent dataset. Statistical evaluations were performed using R software to determine the model's accuracy, sensitivity, specificity, and AUC values. Comparisons with conventional diagnostic methods were conducted to highlight the ThyMPR-CLNM model's advantages.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological confirmation of PTC.
2. Patients who underwent primary surgery accompanied by central neck lymph node dissection.
3. Tumors measuring less than 2 cm in diameter.
4. Postoperative pathological reports including detailed information on the number of lymph nodes dissected and the number of metastatic lymph nodes.
5. Availability of comprehensive preoperative thyroid ultrasound images for analysis.

Exclusion Criteria:

1. Postoperative pathological diagnosis indicating sub-types of PTC.
2. Tumor invasion into adjacent anatomic structures such as the sternothyroid muscle, surrounding soft tissues, trachea, esophagus, or laryngeal nerve.
3. History of neck trauma, previous tumor surgery, or adjuvant chemoradiotherapy.
4. Fewer than three lymph nodes dissected during surgery.
5. Concurrent acute inflammatory conditions or other hematologic disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PTC patients underwent surgery in Hangzhou Traditional Chinese Medical Hospital
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Lymph node metastasis status | Record lymph node metastasis status until the end of the surgery, followed by a one-year follow-up until the conclusion of the study.
  Patients with thyroid cancer undergo thyroid cancer radical surgery according to the guidelines, with pathological results including the number of lymph node metastases and metastasis status, based on the final pathological diagnosis.

SECONDARY OUTCOMES:
Surgical complications and postoperative recurrence | Record surgical complications until the end of the surgery, followed by a one-year follow-up until the conclusion of the study.
  Hemorrhage，Infection，Recurrent laryngeal nerve injury，Hypothyroidism，Other related surgical complications and Recurrence status

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT06725628/Prot_SAP_000.pdf